CLINICAL TRIAL: NCT01698164
Title: Multi-centre Clinical Trial on Hormone Replacement Treatment in China
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008BAI57B04
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Menopausal Syndrome; Cardiovascular Disease; Osteoporosis; Breast Cancer
Keywords: lipid profiles; coronary heart disease; menopausal syndrome; MMSE; MENQOL; HAD
MeSH Terms: conditions — Cardiovascular Diseases; Osteoporosis; Breast Neoplasms; Coronary Disease | interventions — Estradiol; Progesterone

ARMS (3):
- estradiol plus MPA (Active Comparator): 1 mg estradiol valerate, once a day, for 28 days, since the 17th day of taking estradiol valerate adding 4mg medroxyprogesterone acetate, once a day, for 12 days. 28 days forms one cycle. The anticipated duration is 24cycles.
  estradiol valerate, 1mg*21/box medroxyprogesterone acetate, 2mg*100/bottle
  Interventions: Drug: estradiol plus MPA
- estradiol plus progesterone (Experimental): 1 mg estradiol valerate, once a day, for 28 days, since the 17th day of taking estradiol valerate adding 200mg progesterone capsule, once a day, for 12 days. 28 days forms one cycle. The anticipated duration is 24cycles.
  estradiol valerate, 1mg*21/box progesterone capsule, 100mg*6/box
  Interventions: Drug: estradiol plus progesterone
- Ximingting tablet (Experimental): 1 tablet of cimicifuga rhizoma extract, tid 100mg*15*2/box The anticipated duration is 2 years.
  Interventions: Drug: Ximingting Tablet

INTERVENTIONS:
Drug: estradiol plus MPA — Participants are given estradiol and synthetic progestin.
  Arms: estradiol plus MPA
Drug: Ximingting Tablet — Participants are given phytoestrogen.
  Arms: Ximingting tablet
Drug: estradiol plus progesterone — Participants are given estradiol and natural progesterone.
  Arms: estradiol plus progesterone

SUMMARY:
This study is to evaluate the benefit/risk of hormone replacement treatment among early menopausal women in China. This is a multi-centre, random, prospective study.

ELIGIBILITY:
Inclusion Criteria:

* going through amenorrhea above 6 months and within 5 years,
* aged 40 to 60 years,
* going though postmenopausal symptoms,
* serum E2 concentration <30pg/ml,
* serum FSH concentration >40IU/L.

Exclusion Criteria:

* uterine fibroid diameter≥5cm,
* history of diabetes or hypertension,
* history of thromboembolism, severe endometriosis, epilepsy, asthma, hyperprolactinemia,
* first degree relative had a history of breast cancer,
* being in severe or unstable condition of somatic diseases,
* receiving HRT in the past 3 month,
* drug or alcohol abuse in the past 3 month,
* endometrial thickness ≥0.5cm after withdrawal bleeding,
* being allergic to the medicine,
* participating in other clinical trials within 1 month ago.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in risk factors of cardiovascular disease at 12 months and 24 months | before the treatment, time point of taking the medicine for 1 year, time point of taking the medicine for 2 years
  lipid profiles, high-sensitivity C-reactive protein, Hemoglobin A1C, fasting glucose, fasting insulin, blood pressure, waistline, hipline, body composition, electrocardiogram, incidence of coronary heart disease
Change from Baseline in risk factors of breast cancer at 12 months and 24 months | before the treatment, time point of taking the medicine for 1 year, time point of taking the medicien for 2 years
  Mammography, palpation of breast, incidence of breast cancer

SECONDARY OUTCOMES:
Change from Baseline in BMD at 12 months and 24 months | before the treatment, time point of taking the medicine for 1 year, time point of taking the medicien for 2 years
  DEXA bone mineral density
Change from Baseline in risk factors of senile dementia every three months | before the recruitment, before handing out the mecidcine, every three months after taking the medicine till two years later
  mini-mental state examination, hospital anxiety and depression scale
Change from Baseline in the quality of life every three months | before the recruitment, before handing out the mecidcine, every three months after taking the medicine till two years later
  Kupperman menopause index, RAND36 Menopause-Specific quality of life questionaire

OTHER OUTCOMES:
Change from Baseline in thickness of endometrium at 12 months and 24 months | before the treatment, time point of taking the medicine for 1 year, time point of taking the medicien for 2 years
  ultrasonography
uterine bleeding | every three months after taking the medicine until two years later
  diary
Change from Baseline in vital signs every three months | before the recruitment, before handing out the mecidcine, every three months after taking the medicine till two years later
  height, weight, heart rate, BP, gynecological examination
Change from Baseline in general health at 12 months and 24 months | before the treatment, time point of taking the medicine for 1 year, time point of taking the medicien for 2 years
  liver function, renal function

CONTACTS AND LOCATIONS:
Overall Officials: Aijun Sun, PH.D M.D, Study Director — Peking Union Medical College Hospital
Locations (1):
- PUMCH, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xue W, Deng Y, Wang YF, Sun AJ. Effect of Half-dose and Standard-dose Conjugated Equine Estrogens Combined with Natural Progesterone or Dydrogesterone on Components of Metabolic Syndrome in Healthy Postmenopausal Women: A Randomized Controlled Trial. Chin Med J (Engl). 2016 Dec 5;129(23):2773-2779. doi: 10.4103/0366-6999.194646. PMID 27900987